CLINICAL TRIAL: NCT05460507
Title: A Single Arm Open Label Study to Determine the Safety and Efficacy/Tolerability of Rhenium-186 NanoLiposomes (186RNL) for Recurrence of Glioma in Patients Who Received a Prior Treatment With 186RNL
Brief Title: Safety & Efficacy/Tolerability of Rhenium-186 NanoLiposomes (186RNL) for Patients Who Received a Prior 186RNL Treatment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Plus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-GB-001
Record Dates: First submitted 2022-06-13; First posted 2022-07-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Glioma
Keywords: Glioma; Brain Tumor; Radiotherapy; Glioblastoma; Recurrent Glioblastoma; Rhenium; Rhenium Nanoliposome; Brain Cancer; GBM; High Grade Glioma; Glioblastoma Multiform; Grade IV Astrocytoma
MeSH Terms: conditions — Glioma; Brain Neoplasms; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Retreatment with Rhenium Liposome (Experimental): Each participant will receive a single administration of 186RNL. The proposed dose is up to 8.8 mL as a single administration with an administered dose of 22.3 mCi.
  Interventions: Drug: Retreatment Rhenium Liposome

INTERVENTIONS:
Drug: Retreatment Rhenium Liposome — At the time of stereotactic biopsy a catheter will be placed within the tumor using stereotactic guidance. Once the patient has adequately recovered from the procedure as determined by the neurosurgeon, 186RNL will be infused through the CED catheter at the predetermined dose. Spectroscopic imaging will then be obtained at predefined time points to visualize the distribution of the 186RNL as well as calculated the actual dose retained within the tumor. Patients will be monitored longitudinally for evidence of toxicity and response by MRI.
  Other Names: Rhenium-186 NanoLiposome

SUMMARY:
This is an open-label, multicenter, Phase 1 study to establish the safety and efficacy/tolerability of a single dose of 186RNL by the intraventricular route (via intraventricular catheter) for recurrence glioma in patients who received a prior treatment of 186RNL.

DETAILED DESCRIPTION:
This Phase I clinical study evaluates a single dose of 186RNL (radionuclide clinical study drug) administered through a convection enhanced delivery catheter (CED catheter) in participants who have already received a prior treatment of 186RNL.

The clinical study treatment consists of a single administered dose of 186RNL per participant. The proposed dose is up to 8.8 mL as a single administration with an administered dose of 22.3 mCi.

An estimated number of participants to be enrolled in the study is approximately 40.

The clinical study treatment will be administered, following CED placement, by the clinical study physician.

Post-treatment evaluations will be done at Days 3, 7, 14, 28, and every subsequent 28-day interval thereafter until disease progression is confirmed and all treatment related toxicities are resolved. The minimum assessment period for toxicities is 12 weeks.

The U.S. Food and Drug Administration (FDA) has not approved 186RNL for this specific disease.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at time of screening.
2. Ability to understand the purposes and risks of the study and has signed a written informed consent document approved by the site-specific IRB.
3. Patient must present with biopsy and histology proven glioma following initial treatment with 186RNL. The type and grade of glioma to follow the 2021 WHO Classification of Tumors of the Central Nervous System, allowing Grade III and IV gliomas.
4. At least 90 days from prior dose of 186RNL at time of screening.
5. Patients who receive treatment with antiepileptic medications must have a two-week history of stable dose of antiepileptic without seizures prior to dosing.
6. Patients with corticosteroid requirements to control cerebral edema must be maintained at a stable or decreasing dose for a minimum of two weeks without progression of clinical symptoms.
7. A volume of enhancing tumor which falls within the treatment field volume being evaluated in the respective cohort (see 4.1 Design).
8. ECOG performance status of 0 to 2; ECOG 3 acceptable if Principal Investigator and treating physician confirm in patient's interest in study/re-treatment.
9. Life expectancy of at least 2 months
10. Acceptable liver function: Bilirubin ≤ 1.5 times upper limit of normal and AST (SGOT) and ALT (SGPT) ≤ 3.0 times upper limit of normal (ULN)
11. Acceptable renal function: Serum creatinine ≤1.5xULN
12. Acceptable hematologic status (without hematologic support): ANC ≥1000 cells/uL, Platelet count ≥100,000/uL if no bleeding, Hemoglobin ≥7.0 g/dL. Given the absence of hematological toxicity in the ongoing recurrent glioblastoma trial (#12-02) and the need for CED catheter placement, the Investigator and Sub-investigator (neurosurgeon) placing the CED catheter may determine that it is in the patient's best interest and acceptably safe to proceed with this criteria with hematological support or, if no bleeding, Platelet count ≥75,000/uL without support, ANC 1000 cells/uL and Hemoglobin ≥7.0 g/dL
13. All women of childbearing potential must have a negative serum pregnancy test at screening. Male and female subjects must agree to use effective means of contraception (for example, surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose.
14. Patients must have malignant glioma that has progressed on or after standard treatment (surgery, radiotherapy, and/or chemotherapy) and are planned to undergo stereotactic biopsy as per standard of care.

Exclusion Criteria:

1. The subject has evidence of acute intracranial or intratumoral hemorrhage either by MRI or computerized tomography (CT) scan. Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin are eligible.
2. The subject has contraindications to CNS Magnetic Resonance Imaging (MRI).
3. The subject has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for any prior Adverse Events (CTCAE) v4.0 Grade ≤ 1 from AEs (except alopecia, anemia and lymphopenia) due to antineoplastic agents, investigational drugs, or other medications that were administered prior to study.
4. The subject is pregnant or breast-feeding.
5. The subject has serious intercurrent illness, as determined by the treating physician, which would compromise either patient safety include:

   1. Uncontrolled hypertension (two or more blood pressure readings performed at screening of > 150 mmHg systolic or > 100 mmHg diastolic) despite optimal treatment
   2. non-healing wound, ulcer, or bone fracture
   3. clinically significant cardiac arrhythmias affecting cardiac function
   4. untreated hypothyroidism
   5. uncontrolled systemic infection
   6. symptomatic congestive heart failure or unstable, untreated angina pectoris within 3 months prior study drug
   7. myocardial infarction, stroke, transient ischemic attack within 6 months
   8. known active malignancy (other than glioma) except non-melanoma skin cancer or carcinoma in-situ in the cervix
6. The subject has an inherited bleeding diathesis or coagulopathy with the risk of bleeding.
7. The subject has received any of the following prior anticancer therapy:

   1. Non-standard radiation therapy such as brachytherapy, systemic radioisotope therapy, or intra-operative radiotherapy (IORT) to the target site.
   2. Other CNS radiation therapy within 12 weeks of screening.
   3. Systemic therapy (including investigational agents and small-molecule kinase inhibitors) or non-cytotoxic hormonal therapy (e.g., tamoxifen) within 14 days or 5 half-lives, whichever is shorter, prior first dose of study drug
   4. Biologic agents (antibodies, immune modulators, vaccines, cytokines) within 21 days prior to first dose of study drug
   5. Nitrosoureas or mitomycin C within 42 days, or metronomic/protracted low-dose chemotherapy within 14 days, or other cytotoxic chemotherapy within 28 days, prior to first dose of study drug
   6. Prior CNS treatment with carmustine wafers
   7. Patients who are currently receiving any other investigational agents and/or who have received an investigational agent in the prior 28 days from screening.
   8. Patient actively enrolled in an ongoing investigational drug or device trial excluding follow-up only in a previously trial.
8. Multifocal progression or involvement of the leptomeninges.
9. Psychiatric illness/social situations that would limit compliance with the study requirements.
10. Infratentorial disease unless Investigator and neurosurgeon agree it is treated disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of a second dose of 186RNL by CED as part of standard of care >30 days following first dose. | > 30 days
  Safety and tolerability assessed by number of participants with treatment-related toxicities and/or adverse events as assessed by CTCAE v4.0 with 4-week evaluation periods for toxicity and disease assessment until disease progression is suspected.
Overall Survival | 6 Months
  To assess overall survival following 186RNL in patients with bevacizumab naïve recurrent glioblastoma following treatment with a second administration of 186RNL.

SECONDARY OUTCOMES:
Dose Distribution | 3 days
  To assess the dose distribution of a second dose of 186RNL by CED.
Overall Response Rate | 90 days
  To determine the overall response rate by Radiographic Assessment in Neuro-Oncology (RANO) criteria following 186RNL treatment.
Progression-free survival | 6 Months
  To determine disease specific progression-free survival after 186RNL treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Brenner, PhD, Principal Investigator — The Cancer Therapy and Research Center at UTHSCSA
Locations (1):
- The Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No